CLINICAL TRIAL: NCT02552693
Title: Enhancing Retention in Care for HIV-positive Mothers and Their Infants by Improving Facility Tracking and Community Health Worker Tracing in Zimbabwe
Brief Title: The TracTOR (Tracking and Tracing Operations Research) Study -- Zimbabwe
Acronym: TracTOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elizabeth Glaser Pediatric AIDS Foundation (Other)
Collaborators: Population Council (Other)
Responsible Party: Principal Investigator, Godfrey Woelk, Director of Global Implementation Research, Elizabeth Glaser Pediatric AIDS Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EG0137
Record Dates: First submitted 2015-09-15; First posted 2015-09-17 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: HIV
Keywords: Enhancing retention
MeSH Terms: interventions — Organization and Administration; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Facility (Experimental): Enhanced training, supervision and support for MOHCC Standard Operating Procedure (SOP) implementation of identifying, tracing and returning to care (tracking and tracing) defaulting mother/infant pairs.
  Facilities in the experimental group will receive additional training, supervision and support in identifying, tracing and returning to care defaulting mother/infant pairs.
  Interventions: Other: Enhanced training, supervision and support
- Control Facility (No Intervention): Facilities in the control group will be operating as described in the MOHCC SOP. (Standard practice in tracking and tracing of defaulting mother/infant pairs)

INTERVENTIONS:
Other: Enhanced training, supervision and support — The intervention includes the following activities:
  Conduct of pre-intervention facility audits; Cross-verification of appointment diaries with facility attendance records; Development and implementation of job aids and tools; Provides supplemental training and technical support to focal facility point (FFP) and other staff, and community health workers (CHWs); Improves coordination, supervision and reporting systems at the health facilities.
  Arms: Experimental Facility

SUMMARY:
This study evaluates the effectiveness of an enhanced package of support for activities described in the "Standard Operating Procedures (SOP) for Patient Tracing in Health Facilities in Zimbabwe". This package is intended to increase the effectiveness of active patient tracing activities by developing tools, providing mentorship and implementing systematic review of processes to improve communication, coordination, and supervision between community health workers and facility-based staff.

DETAILED DESCRIPTION:
This study consists of a pre-/post- intervention rapid assessment of SOP implementation in study health facilities. The rapid assessment includes a facility audit, and the cross-verification of Mother-baby pair service records, and scheduled appointments. Following the baseline rapid assessment, the research team implements the proposed intervention package in health facilities randomly assigned to the intervention arm of the study. Data collectors conduct monthly visits to study facilities in order to extract appointment attendance information from PMTCT, ART, pharmacy, HIV exposed infants (HEI), and early infant diagnoses (EID) service registers.

ELIGIBILITY:
Inclusion Criteria:

Mother-baby pair (MBP):

1. Mother is HIV-positive
2. Infant was born between October 1st, 2013 and March 30th, 2015, or initiates HIV exposed infant services within the first seven months of the data collection period
3. Mothers and infants are assigned unique facility-issued ID numbers that can be used to pair their records, and link service attendance between clinical units, and over time
4. Enrolled in post-natal PMTCT, ART, or EID services at a study health facility
5. Based on guidelines in the SOP, MBP cannot be classified as lost to follow-up at beginning of data collection period

Community Health Workers (CHW):

1. CHW or facility-based staff working at selected study sites
2. Participated in the implementation of MBP tracking and tracing activities for a minimum of three months
3. Participant in district-level or selected facility-level CHW meetings
4. Above age of consent (18 years or above)
5. Able and willing to provide informed consent to participate in the study

Exclusion Criteria:

* If inclusion criteria not met

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 946 (Actual)
Dates: Start 2015-03; Primary Completion 2016-03 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Proportion of HIV positive women traced | 6 months
  To determine whether the strategies proposed to enhance support for the implementation of Zimbabwe's patient tracing SOP affect rates of MBP retention in PMTCT programs, and infant HIV testing.

SECONDARY OUTCOMES:
Proportion of HIV exposed infants tested for HIV | 6 months
  To document the implementation of mother-baby-pair tracking and tracing activities; and assess their fidelity to the SOP.

CONTACTS AND LOCATIONS:
Overall Officials: Godfrey B Woelk, PhD, Principal Investigator — Elizabeth Glaser Pediatric AIDS Foundation
Locations (1):
- EGPAF Zimbabwe, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
Dataset has been shared with the USAID study sponsor who will make data available in 2018